CLINICAL TRIAL: NCT05144958
Title: Stand-Alone Left Atrial Appendage Occlusion for throMboembolism Prevention in Nonvalvular Atrial fibrillatioN DiseasE Registry (SALAMANDER)
Brief Title: Stand-alone Left Atrial Appendage Occlusion for Thromboembolism Prevention
Acronym: SALAMANDER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Mariusz Kowalewski, PhD, M.D., Nicolaus Copernicus University
Other Study IDs: SALAMANDER
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Totally thoracoscopic LAAO - ATRICLIP: In this group, LAA will be sealed using the epicardial thoracoscopic approach with the ATRICLIP device.
  Interventions: Device: Totally thoracoscopic LAAO - ATRICLIP
- Percutaneous LAAO - WATCHMAN: In this population, LAA will be occluded using an endocardial totally-percutaneous approach with the WATCHMAN device.
  Interventions: Device: Percutaneous LAAO - WATCHMAN
- Hybrid- minimally invasive LAAO - LARIAT: In these patients, LAA will be closed using a hybrid, combined endo- and epicardial approach using the LARIAT system.
  Interventions: Device: Hybrid- minimally invasive LAAO - LARIAT

INTERVENTIONS:
Device: Totally thoracoscopic LAAO - ATRICLIP — The device for surgical totally thoracoscopic left atrial appendage occlusion AtriClip® Gillinov-Cosgrove™ (AtriClip, AtriCure, Dayton, OH, USA) consists of an automatically closing clip placed in a deployment loop on a disposable holder with the head articulation of 60 degrees side-to-side and up/down. The several novel features of the system in comparison to previous ones, such as its length, maneuverability and releasing system, enable it to be used in a totally thoracoscopic fashion. The AtriClip® PRO has parallel titanium crossbars that equalize the force over the tissue trabeculations of the LAA during deployment, ensuring a sealed line at the base of the LAA orifice, as confirmed in preclinical and clinical studies. The clip can be opened and closed repeatedly before final deployment when only the correct placement is confirmed in TEE.
  Groups: Totally thoracoscopic LAAO - ATRICLIP
Device: Percutaneous LAAO - WATCHMAN — Using a modified Seldinger technique a vessel dilator and a guidewire are inserted into the femoral vein. Under trans-esophageal echocardiography and fluoroscopy guidance, an interatrial septum is punctured using typical trans-septal access. The pigtail catheter is placed in the distal portion of the left atrial appendage and then the access sheath is inserted. After choosing the appropriate Watchman size the device is deployed and seals the left atrial appendage.
  Groups: Percutaneous LAAO - WATCHMAN
Device: Hybrid- minimally invasive LAAO - LARIAT — LARIAT system consists of: A) endocardial magnet-tipped guidewire. It is placed inside the left atrial appendage through the introduction of a catheter into the femoral vein; B) epicardial magnet-tipped guidewire. It is placed on the outside of the left atrium through the atrial appendage puncture of the pericardium. Each wire has a magnet of opposite polarity enabling end-to-end alignment; C) A compliant occlusion balloon catheter to identify the LAA and allow for a very precise and effective seal of the left atrial appendage; D) The LARIAT suture delivery device. It is introduced by an earlier puncture of the pericardium in the vicinity of the left atrial appendage and guided over magnet wire onto the base of the LAAO. With the LARIAT suture delivery device, the lumen of the left atrial appendage is closed from outside the heart, resulting in the elimination of the thrombus source.
  Groups: Hybrid- minimally invasive LAAO - LARIAT

SUMMARY:
This prospective nationwide registry aims to assess the durability of left atrial appendage occlusion when performed via totally thoracoscopic, percutaneous and hybrid- minimally invasive approaches and collect information on possible adverse events.

DETAILED DESCRIPTION:
Stand-Alone Left Atrial appendage occlusion for throMboembolism prevention in Nonvalvular Atrial Fibrillation DiseasE Registry (SALAMANDER) will commence in 37 heart surgery centers across Poland and has no limit of patient recruitment. Included in the registry will be all >18 y.o. patients with AF and high risk of thromboembolic and bleeding complications defined by CHA2DS2-VASc Score > 2 and HASBLED score of > 2 referred to stroke prevention who do not require an open chest surgery for other reasons. The primary outcome will be the number of perioperative (in-hospital/30-days) complications associated with LAA closure device placement and intraoperative success of exclusion of LAA as assessed by transesophageal echocardiography. Secondary outcomes will be major adverse cardiac and cerebrovascular events (MACCE, combined endpoint of death, acute heart failure, myocardial infarction and stroke); pulmonary complications and any complications connected with surgical intervention. AF-related risks, including stroke/systemic thromboembolism and bleeding outcomes, will be assessed. Medical history, risk factors, demographic information and management will be collected at baseline, and clinical events during 1 -year follow-up will be recorded. Follow-up will be conducted for at least 1 year and then annually thereafter till year 5th post-op.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged ≥18 years;
2. ECG/Holter diagnosis of AF;
3. Previous stroke or systemic thromboembolic complications;
4. High risk of thromboembolic complications - CHA2DS2-VASc Score ≥ 2;
5. HASBLED score of > 2;
6. Contraindications to oral anticoagulation or Complications of oral anticoagulation;

(8) Acceptable surgical candidate, including use of general anesthesia; (9) patient adherence to the study and patient Informed Consent Form has been signed

Exclusion Criteria:

1. No ECG with AF recorded (12-lead ECG, Holter recording, external event recorder or implantable loop recorder) or only atrial flutter recorded,
2. Significant valve disease or coronary multivessel artery lesions requiring operation;
3. Stroke/cerebrovascular accident (CVA) within previous 30 days;
4. Critical preoperative state;
5. participation in a clinical trial
6. patient refusal

Registry imposes intraoperative exclusion criteria to otherwise enrolled patients:

1. Presence of thrombus in the LA or LAA
2. LAA tissue with significant adhesions (as evaluated by the surgeon) making AtriClip® placement overly risky.
3. Previous cardiac operations (e.g., CABG, heart transplant, valvular replacement) making LARIAT placement overly risky.
4. Patients with a previous atrial septal defect with surgical or transcatheter closure making Watchman placement overly risky.
5. NYHA IV;
6. Right-sided heart failure;
7. Symptomatic carotid artery disease;
8. active systemic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-valvular AF and high risk of thromboembolic and bleeding complications defined by CHA2DS2-VASc Score > 2 and HAS-BLED score of > 2 referred to stroke prevention who do not require an open chest surgery for other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy | 30 days
  The number of peri-operative (in-hospital/30-days) complications associated with LAA closure device placement and intraoperative success of exclusion of LAA as assessed by transesophageal echocardiography

SECONDARY OUTCOMES:
Long-term sequelae | 5 years
  Major adverse cardiac and cerebrovascular events (MACCE, combined endpoint of death, acute heart failure, myocardial infarction and stroke); pulmonary complications and any complications connected with surgical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiac Surgery, Centre of Postgraduate Education, Warsaw, Mazovian, Poland

REFERENCES:
- [Derived] Kowalewski M, Wanha W, Litwinowicz R, Kolodziejczak M, Pasierski M, Januszek R, Kuzma L, Grygier M, Lesiak M, Kaplon-Cieslicka A, Reczuch K, Gil R, Pawlowski T, Bartus K, Dobrzycki S, Lorusso R, Bartus S, Deja MA, Smolka G, Wojakowski W, Suwalski P. Stand-Alone Left Atrial appendage occlusion for throMboembolism prevention in nonvalvular Atrial fibrillatioN DiseasE Registry (SALAMANDER): protocol for a prospective observational nationwide study. BMJ Open. 2022 Sep 21;12(9):e063990. doi: 10.1136/bmjopen-2022-063990. PMID 36130748